CLINICAL TRIAL: NCT02922556
Title: Piloting a Novel, Mobile Cognitive Training Tool for Patients With Major Depressive Disorder (MDD)
Acronym: MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1008-2015
Record Dates: First submitted 2016-07-13; First posted 2016-10-04 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Games, Experimental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training (Moodify) requiring a total maximum of 50 treatment hours, 3-5 times weekly, 30-45 minutes each session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training (Games) requiring a total maximum of 50 treatment hours, 3-5 times weekly, 30-45 minutes each session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Other Names: Moodify
  Arms: Experimental Treatment
Other: Commercially available computerized training
  Other Names: Games
  Arms: Active Comparator

SUMMARY:
To assess the efficacy of a mobile-device-deployed cognitive emotional treatment for depression (Moodify) versus an active control treatment (commercially available computer games).

DETAILED DESCRIPTION:
The study will involve a randomized, controlled, double-blind trial to assess the efficacy of a mobile-device-deployed cognitive emotional treatment for depression (Moodify) versus an active control treatment (commercially available computer games). Moodify is comprised of a novel continuous performance task (CPT) to improve cognitive slowing and lethargy often present in cases of major depressive disorder. This training method is based on an existing, validated cognitive training paradigm (tonic and phasic attention training, TAPAT1; WIRB Study No. 1126399). Moodify will also employ two additional cognitive training modules previously validated in this and other clinical populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants must 18 to 85 years or older and not pregnant
* Participants must be fluent in English
* Participants must be able to engage with computerized cognitive tasks as required in order to participate in this study.
* Normal vision (or corrected to normal vision)
* Participants must be willing to commit to the time requirements of the study as evidenced by written, informed consent.
* Participants must meet diagnostic criteria for MDD

Exclusion Criteria:

* Participants report or present a hand tremor that prevents the use of a computer mouse or keyboard
* Participants unable to perform neuropsychological evaluations
* Participants cannot comprehend or follow instructions
* Participants not capable of giving informed consent
* Participants who appear to be intoxicated or under the influence of a controlled substance
* Participants with a history of significant medical diseases or multiple neurological events of the head
* Participants with serious or unstable medical illness (e.g. cardiovascular, hepatic, renal, endocrine, neurologic disease)
* Participants with a history or current diagnosis to specific Diagnostic and Statistical Manual (DSM)-IV psychiatric illness such as (but not limited to): organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder Not Otherwise Specific, bipolar disorder, substance dependence and substance abuse
* Participants with a history of seizure disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change scores for depressive symptoms using Beck Depression Scale (BDI) | 3 months and 6 months
Change scores for anxiety symptoms using Generalized Anxiety Disorder (GAD-7) | 3 months and 6 months
Change scores for functional health and well being using the 12-Item Short Form Health Survey (SF-12) | 3 months and 6 months
Change scores for depressive symptoms using Patient Health Questionnaire (PHQ-9) | 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Posit Science Corporation, San Francisco, California, United States